CLINICAL TRIAL: NCT07092592
Title: Developing an Optical Coherence Tomography (OCT) Based Handheld Intraoral Scanner for Dentistry
Brief Title: Optical Coherence Tomography (OCT) Based Intraoral Scanner
Status: Not yet recruiting | Type: Observational
Sponsor: Perceptive Technologies, Inc (Industry)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); The Forsyth Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PerceptiveTech; 1R44DE033316 (NIH)
Record Dates: First submitted 2025-06-16; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: The Focus of the Study is to Evaluate the Efficacy of OCT in Scanning and Reconstructing General Tooth and Gum Anatomy; Tooth Anatomy; Gingival Anatomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to optimize the matching between Optical Coherence Tomography (OCT) imaging and the true anatomy of the tooth. It also non-invasively tests how reliable the OCT scanner can access tissue integrity, measure depth, and detect texture features. These features will be important to plan for treatment. The specific aims of this study are:

1. to correct for distortion caused by internal refractive indices to restore true tooth anatomy
2. to test the feasibility and usability of the full-motion OCT scanner in volunteers.

Participants may be in one of the following groups

1. Some teeth that are extracted according standard treatment plan will be scanned with OCT.
2. Some participants will have their teeth and gum in the mouths scanned by OCT

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to agree by the terms of the consent form and sign the Informed Consent form
* Aged 18 years old and older
* Individuals with a minimum of 18 natural teeth present including teeth from distinct groups (molar, premolar and anterior teeth).
* Having healthy dentition (small carious lesions and dental restorations not covering the entire surface of the tooth will be accepted) as determined by the dental clinician
* Willing to have a retraction cord placed under the gumline for a duration of 2 min.
* Having a tooth that requires crown procedure according to treatment planning by the patients' clinician (for real-time scanning)

Exclusion Criteria:

* Pregnant women
* Generalized gingivitis and periodontal disease
* Extensive dental work including dental fillings, crowns and implants and extensive tooth damage (i.e., fracture, large dental caries, etc.)
* Presence of fixed orthodontic braces, or lingual bars (only for in vivo studies)
* Presence of generalized (or on target teeth) supra and subgingival calculus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All study participants will be recruited at the Forsyth Center for Clinical and Translational Research and Forsyth Faculty Associates Clinics (those scheduled for tooth extractions). Potentially eligible participants will be invited to the initial screening visit, in which they will be asked to complete medical and dental history, and will undergo a clinical examination. After selection of those who fulfill the inclusion and exclusion criteria, study participants will be provided with details of the trial.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-08-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Intra-method reliability/repeatability testing | Up to 24 weeks
  Intra-class correlation coefficients will be calculated for tissue characteristics listed above will be determined by the OCT scanner on group of teeth (full-arch), single tooth and subgingival surfaces.

SECONDARY OUTCOMES:
Structure assessments | Up to 24 weeks
  Extracted teeth will be scanned with the OCT scanner. The air-enamel interface and the internal structure (e.g. Dentin-Enamel Junction) will be detected in the OCT reconstructed images. The ground truth of the anatomy will be provided by histology or micro-CT. The OCT reconstructed anatomy will be compared to the ground truth to understand the accuracy of the OCT scanner.

CONTACTS AND LOCATIONS:
Locations (1):
- The ADA Forsyth Institute, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The IPD will be for internal use only.